CLINICAL TRIAL: NCT00614562
Title: Neurally Adjusted Ventilatory Assist (NAVA) in Patients With Critical Illness Associated Polyneuropathy / or Polymyopathy (CIP/M)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Lukas Brander, MD, University Hospital - Inselspital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KEK BE 250/07
Record Dates: First submitted 2008-01-31; First posted 2008-02-13 (Estimated); Last update posted 2011-02-03 (Estimated); Status verified 2011-02

CONDITIONS: Polyneuropathy; Polymyopathy
Keywords: critical associated illness polyneuropathy or polymyopathy (CIP/M)
MeSH Terms: conditions — Polyneuropathies | interventions — Interactive Ventilatory Support

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- NAVA (Experimental)
  Interventions: Device: Neurally adjusted ventilatory assist (NAVA)

INTERVENTIONS:
Device: Neurally adjusted ventilatory assist (NAVA) — NAVA for 72 hours

SUMMARY:
Neurally adjusted ventilatory assist (NAVA) is a new concept of mechanical ventilation. NAVA delivers assist to spontaneous breathing based on the detection of the electrical activity of the diaphragm. We study the effect of NAVA in patients with critical illness associated polyneuropathy / polymyopathy (CIP/M)

ELIGIBILITY:
Inclusion Criteria:

1. Subject itself or its next of kin has given written informed consent
2. Independent physician has given written informed consent
3. Male or female patients aged 18 - 80 years (extremes included).
4. Mechanical ventilation for ≥ 48 hours prior to enrolment
5. Presence of Critical Illness Polyneuropathy / Polymyopathy (CIP/M) according to the MRC Scale for Muscle Examination in 12 Muscle groups (Table 1) with or without loss of sensibility and muscle reflexes.
6. Presence of at least one of the following risk factors (A - D) known to be associated with CIP/M. Note, the risk factor does not need to be present at enrolment but needs to have been present prior to enrolment during the actual stay in the ICU:

   * A: severe sepsis defined as the presence of an infection is highly suspected or proven and three or more of the following systemic inflammatory response syndrome (SIRS) criteria are met (Bernard et al 2001 s. Figure 15):

     * core temperature greater than 38 degrees celsius (100.4 degrees F) or less than 36 degrees celsius (96.8 degrees F);
     * heart rate greater than 90 beats per minute;
     * respiratory rate greater than 20 breaths per minute, or arterial carbon dioxide tension (Paco2) greater than 32 mm Hg, or mechanical ventilation for an acute process;
     * a white cell count of more than 12 000/mm3 or less than 4000/mm3 , or a differential count showing more than 10% immature neutrophils.
   * B: MODS (s. Figure 15)
   * C: treatment with corticosteroids for at least 24 hours (either as repeated bolus or as continuous infusion).
   * D: treatment with neuro-muscular blocking agents for at least 24 hours (either as repeated bolus or as continuous infusion).

Exclusion Criteria:

1. Patient is less than 18 years or more than 80 years of age
2. The attending physician refuses to allow enrollment
3. The patient refuses informed consent
4. Next of kin is unavailable or refuses informed consent
5. The independent physician refuses informed consent
6. Pregnant or breast-feeding female. A pregnancy test will be performed in all female patients less than 60 years of age
7. Any contraindication to insertion/exchange a nasogastric tube, including (but not limited to): severe oropharyngeal malformation or bleeding; esophageal varices, tumor, infection, stenosis, or rupture, bleeding disorder with evidence of active bleeding.
8. Presence or suspicion of diaphragm injury
9. Presence or suspicion of a central nervous system (CNS) proximal of the spinal cord level C2) including (but not limited to): infarction, bleeding, tumor, or infection in the CNS
10. Presence or suspicion of any preexisting peripheral neuromuscular disorder.
11. History of heart and/or lung transplantation
12. Any mechanical cardiac assist device (excluding intraaortic balloon pump)
13. Any contraindication to reduce sedation or to stop neuromuscular blockage in order to allow spontaneous breathing
14. The patient needs to be ventilated with a mode of mechanical ventilation that targets a redefined tidal volume or airway pressure as per attending physician
15. Severe hemodynamic instability as per attending physician
16. A fraction of inspired oxygen (FiO2) of > 0.8 at enrollment.
17. The patient currently participates in another interventional clinical trial

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2008-01; Primary Completion 2009-06 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Changes in mean inspiratory electrical activity of the diaphragm (Edi) | beginning to end of study

SECONDARY OUTCOMES:
Changes in ventilatory and respiratory parameters Changes in sedative and vasoactive drugs used | beginning to end of study

CONTACTS AND LOCATIONS:
Overall Officials: Lukas Brander, MD, Principal Investigator — Department of Intensive Care Medicine, University Hospital, Bern, Switzerland
Locations (1):
- Department of Intensive Care Medicine, University Hospital - Inselspital, Bern, Switzerland

REFERENCES:
- [Background] Sinderby C, Navalesi P, Beck J, Skrobik Y, Comtois N, Friberg S, Gottfried SB, Lindstrom L. Neural control of mechanical ventilation in respiratory failure. Nat Med. 1999 Dec;5(12):1433-6. doi: 10.1038/71012. No abstract available. PMID 10581089
- [Derived] Tuchscherer D, Z'graggen WJ, Passath C, Takala J, Sinderby C, Brander L. Neurally adjusted ventilatory assist in patients with critical illness-associated polyneuromyopathy. Intensive Care Med. 2011 Dec;37(12):1951-61. doi: 10.1007/s00134-011-2376-0. Epub 2011 Nov 3. PMID 22048718